CLINICAL TRIAL: NCT01842464
Title: Sacro-Spinous Ligaments Anterior Apical Anchoring for Needle-Guided Mesh in Advanced Pelvic Organ Prolapse
Brief Title: Sacro-Spinous Ligaments Anterior Apical Anchoring
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, menahem neuman, Responsible for UroGynecology and Pelvic Floor Medicine, Western Galilee Hospital-Nahariya
Other Study IDs: WesternGalileeH
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Anterior Sacro-Spinous Support: Anterior sacro-spinous mesh implants supported patients
  Interventions: Procedure: Anterior Sacro-Spinous

INTERVENTIONS:
Procedure: Anterior Sacro-Spinous — Anterior Sacro-Spinous

SUMMARY:
Anterior-apical compartment mesh implants for pelvic floor reconstruction are anchored here to the Sacro-Spinous ligaments and evaluated being a feasible and effective method.

DETAILED DESCRIPTION:
Anterior-apical compartment mesh implants for pelvic floor reconstruction are frequently anchored to the Arcus Tendinous Fascia Pelvis (ATFP) rather than to the Sacro-Spinous (SS) ligaments commonly used for the posterior compartment reconstruction. The SS ligament suspension for apical support mesh fixation is thought to yield higher and stronger anchoring point than the ATFP. The authors presumed that anterior mesh fixation to the sacro-spinous ligament are both, feasible and effective.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic Floor Prolapse > Gr 2,
* Anterior > Posterior defect,
* Apical Supportive Defect

Exclusion Criteria:

* Active Pelvic Inflammation,
* Patient Refusal

Ages: 35 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients suffering advanced pelvic organ prolapse with anterior predominance and apical supportive defect, reffered to mesh reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Menahem Neuman, Prof., Principal Investigator — Western Galilee MC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 patients with significant Pelvic Organ Prolapse requiring mesh reconstruction during 2011-2012
Pre-assignment Details: The study patients were retrieved out of the operated patients population during the study period.
Groups:
- Anterior Sacro-Spinos Support: Anterior Sacro-Spinous Support :
Period: Overall Study
Arm/Group | Anterior Sacro-Spinos Support
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anterior Sacro-Spinos Support
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change With Distance Between the Vaginal Apex and the Introitus
Description: The change with distance measured by centimeters, between the vaginal apex and the introitus
Time Frame: One year
Measure: Mean (Full Range); unit: centimeters
Groups:
- Anterior Sacro-Spinous Support: Number of participants with successful Sacro-Spinous Ligaments Anterior Apical Anchoring
Arm/Group | Anterior Sacro-Spinous Support
Number analyzed (Participants) | 44
centimeters | -4.4 [-7 to 7]

2. Primary Outcome: Efficacy of Sacro-Spinous Ligaments Anterior Apical Anchoring
Description: Level of support with the Sacro-Spinous Ligaments Anterior Apical Anchoring higher than 4 centimeters above vaginal opening.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Anterior Sacro-Spinos Support
Number analyzed (Participants) | 44
participants | 44

3. Primary Outcome: Number of Participants Involving in Complications: Operative Damage and Bleeding, Post Operative Infection and Mesh Exposure
Description: Number of participants involving in complications: operative damage and bleeding, post operative infection and mesh exposure.
Time Frame: one year
Population: occurrence and severity of complication is recorded
Measure: Number; unit: participants
Arm/Group | Anterior Sacro-Spinos Support
Number analyzed (Participants) | 44
participants | 0

ADVERSE EVENTS:
Time Frame: one year
Description: Urinary tract injury, intestinal injury, nerve injury, bleeding, mesh exposure, infection,
Arm/Group | Anterior Sacro-Spinos Support
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No